CLINICAL TRIAL: NCT00782028
Title: Integrating Well-Woman and Well-Baby Care to Improve Parenting and Family Wellness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: John M. Leventhal, MD, Department of Pediatrics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R21 HDJ2810-01A1
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Primary Care
Keywords: primary care, high-risk families, maternal depression
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): No intervention consists of routine well child care
  Interventions: Other: Standard Care
- Centering parenting/Group well child care (Other)
  Interventions: Other: Centering parenting/Group well child care

INTERVENTIONS:
Other: Centering parenting/Group well child care — Intervention families will receive well child care in a group format for the first 12 month of the child's life.
  Arms: Centering parenting/Group well child care
Other: Standard Care
  Arms: Standard Care

SUMMARY:
We hypothesize that relative to families who receive standard individual postpartum and pediatric care, families that receive group care will be more likely to have:

* Improved maternal and child health behaviors: i.e increased breastfeeding, exercise, child safety measures in the home and decreased smoking.
* Better health care use for babies: i.e. attend more care visits, on-time and complete immunizations and decreased emergency services use.
* Better psychosocial outcomes for the families: i.e. decreased stress and depression, and increased social support.
* Improved parenting skills: i.e. improved knowledge of child development, involvement in developmentally appropriate activities, and parental sense of competence.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum woman with baby in her care
* Receive well-woman care, well-child care and interviews in English
* Willingness to receive care in a group setting
* Woman planning to receive care at the Yale Women's Center for herself and the Primary Care Center for her baby

Exclusion Criteria:

* severe medical problem requiring individualized care for mother or baby
* Baby born at less than 37 weeks gestation
* Baby remaining in hospital when mother getting discharged for any other reason except hyperbilirubinemia
* Baby with severe cardiac, respiratory, neuro-developmental or surgical problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Improved maternal and child health behaviors will be measured using a computer assisted interview. | Interviews will be given at 2 weeks, 6 and 12 months of age.

SECONDARY OUTCOMES:
Better health care utilization for babies will be measured using Medical records review. | 1 year
Better psychosocial outcomes for mothers, fathers and babies will be measured using a computer assisted interview. | 2 weeks, 6 months and 12 months of age
Improved parenting skills will be assessed using a computer assisted inteview. | 2 weeks, 6 months ad 12 months